CLINICAL TRIAL: NCT04796259
Title: Malt-derived Ingredients and Their Prolactinotrophic Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20.21.NRC
Record Dates: First submitted 2021-03-11; First posted 2021-03-12 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Acute Response to Food Ingredient Consumption

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Negative control (No Intervention): Water
- Positive control (Active Comparator): Non-alcoholic beer solids
  Interventions: Dietary Supplement: Non-alcoholic beer solids
- Intervention 1 (Experimental): Malt ingredient I
  Interventions: Dietary Supplement: Malt ingredient
- Intervention 2 (Experimental): Malt ingredient II
  Interventions: Dietary Supplement: Malt ingredient

INTERVENTIONS:
Dietary Supplement: Malt ingredient — Solution with malt-derived ingredient
  Arms: Intervention 1; Intervention 2
Dietary Supplement: Non-alcoholic beer solids — Solution with non-alcoholic beer solids
  Arms: Positive control

SUMMARY:
This proof-of-concept study aims to investigate whether malt-derived ingredients have acute prolactinotrophic effects in healthy women of child-bearing age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have/are

  1. Willing and able to provide written informed consent
  2. Healthy women aged 18 to 40.
  3. BMI in the range of 18 to 30.
  4. Willing to undergo an experiment in the follicular phase of the menstrual cycle i.e. day 0 to 14 of the menstrual cycle starting from the first day of the period.

Exclusion Criteria:

* Subjects who have/are
* Allergic to tested products
* Under regular medication including oral contraceptive pills or other form of hormonal replacement therapy.
* Under medications which affects prolactin levels.
* Pregnant or lactating or planning to conceive during the study period.
* Smokers, or excessive alcohol consumption (alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer) or other substance abuse.
* Not willing and/or not able to comply with the study procedures and requirements.
* Suffering from pre-existing medical conditions and chronic illnesses that in the opinion of the investigator may interfere with the study.
* Family or hierarchical relationships with research team members

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Prolactinotrophic effect | 2 hours post consumption
  Δ of serum Prolactin Cmax between test products, positive control of beer solids and negative control of still water

SECONDARY OUTCOMES:
Gastrointestinal tolerability | 2 hours post consumption
  • Gastro-intestinal tolerability assessment with a visual analogue scale for each symptom of interest i.e.1) Abdominal discomfort 2) Nausea 3) Vomiting 4) Diarrhoea 5) ↓appetite.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M. Ramos Nieves, M.Sc.; Ph.D., Principal Investigator — Société des Produits Nestlé S.A./NIHS; Pamela Sun, Study Director — Société des Produits Nestlé S.A./CIL
Locations (1):
- Société des produits Nestlé/Metabolic Unit, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No